CLINICAL TRIAL: NCT00274677
Title: A Multicenter, Double-Blind, Placebo-Controlled, Fixed-Dose, 8-Week Evaluation of the Efficacy and Safety of Lamotrigine in the Treatment of Depression in Patients With Type II Bipolar Disorder
Brief Title: Depression And Bipolar Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCA100223; NCT00076882 (obsolete NCT alias)
Record Dates: First submitted 2006-01-09; First posted 2006-01-11 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Bipolar Disorder
Keywords: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Lamotrigine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: lamotrigine
- lamotrigine (Experimental)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Experimental treatment arm
  Arms: lamotrigine
Drug: lamotrigine — Experimental treatment
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
This study is an 8-week evaluation of an investigational drug for treating depression in bipolar patients. Depressed patients will be given either an investigational drug or placebo and receive psychiatric assessments of their depression at weekly visits. Study drug and all study-related visits are provided at no cost to the patient. The patient agrees to meet with study research staff for roughly 11 clinic visits.

ELIGIBILITY:
Inclusion

* Patients must provide written and informed consent.
* Diagnosis of Bipolar II Disorder and currently depressed for minimum of the last 8 weeks.

Exclusion

* Patients must not be suicidal.
* Patients must not have a history of non-response to antidepressant treatment.
* Patients must not have a clinical history of substance dependence in the past year or abuse within the 4 weeks prior to study entry.
* Patients must not have had epilepsy or hypothyroidism.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2003-11; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline scores at Week 8 for the Montgomery-Asberg Depression Rating Scale (MADRS) | Eight weeks

SECONDARY OUTCOMES:
Change from baseline scores at Week 8 for the Hamilton Depression Rating Scale (HAMD-17, HAMD-31, Bech Melancholia Scale (BMS), and HAMD (Item 1), Clinical Global Impressions of Severity (CGI-S) and Improvement (CGI-I) | Eight weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (19):
- United States (19):
  - GSK Investigational Site, Burbank, California
  - GSK Investigational Site, Loma Linda, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Marietta, Georgia
  - GSK Investigational Site, Terre Haute, Indiana
  - GSK Investigational Site, Shreveport, Louisiana
  - GSK Investigational Site, Saint Charles, Missouri
  - GSK Investigational Site, Clementon, New Jersey
  - GSK Investigational Site, Princeton, New Jersey
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Pleasantville, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Beachwood, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Eugene, Oregon
  - GSK Investigational Site, Columbia, South Carolina
  - GSK Investigational Site, Galveston, Texas
  - GSK Investigational Site, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Hashimoto Y, Kotake K, Watanabe N, Fujiwara T, Sakamoto S. Lamotrigine in the maintenance treatment of bipolar disorder. Cochrane Database Syst Rev. 2021 Sep 15;9(9):CD013575. doi: 10.1002/14651858.CD013575.pub2. PMID 34523118
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: SCA100223 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: SCA100223 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: SCA100223 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: SCA100223 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: SCA100223 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: SCA100223 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: SCA100223 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register